CLINICAL TRIAL: NCT05745623
Title: A Multi-center, Non-Randomized, Open-Label Phase 2 Basket Clinical Trial to Evaluate ICP-723 in Patients With Advanced Solid Tumors or Primary Central Nervous System Tumors
Brief Title: Study of ICP-723 in Patients With Advanced Solid Tumors or Primary Central Nervous System Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00505
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors Harboring NTRK Fusion; Primary Central Nervous System Tumors Harboring NTRK Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICP-723 (Experimental)
  Interventions: Drug: ICP-723

INTERVENTIONS:
Drug: ICP-723 — ICP-723 tablet administered orally，once a day，for every 28 days as one cycle

SUMMARY:
A Multi-center, Non-Randomized, Open-Label Phase 2 Basket Clinical Trial to Evaluate ICP-723 in Patients with Advanced Solid Tumors or Primary Central Nervous System Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
2. Patients with advanced solid tumors or primary central nervous system (CNS) tumors harboring NTRK gene fusions as detected by the designated central laboratory, who received no previous NTRK inhibitor treatment;
3. At least one measurable lesion as per RECIST1.1 criteria, or for primary CNS tumors, at least one measurable lesion as per RANO or INRC criteria.
4. Organ functions meet the clinical criteria

Exclusion Criteria:

1. Patients with unstable primary central nervous system (CNS) tumors or CNS metastasis.
2. Patients with abnormal QTc interval at screening, or other clinically significant abnormalities in electrocardiographic examination at the discretion of the investigator.
3. Patient with recent anti-tumor and other treatment as stated in the protocol.
4. Grade 1 or higher toxicities attributed to any previous treatment not yet recovered.
5. Other conditions considered unsuitable for participation in this trial at the discretion of the investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 4 years
  The objective response rate (ORR) evaluated by the Independent Center Review

SECONDARY OUTCOMES:
ORR assessed by the investigator | Through study completion, an average of 4 years
DCR as assessed by the investigator and the IRC | Through study completion, an average of 4 years
Time to response (TTR) as assessed by the investigator and the IRC | Through study completion, an average of 4 years
Duration of response (DOR) as assessed by the investigator and the IRC | Through study completion, an average of 4 years
Progression-free survival (PFS) as assessed by the investigator and the IRC | Through study completion, an average of 4 years
Intracranial objective response rate (IC-ORR) as assessed by the investigator and IRC | Through study completion, an average of 4 years
central nervous system progression-free survival (CNS-PFS) as assessed by the investigator and IRC | Through study completion, an average of 4 years
Overall survival (OS) | Through study completion, an average of 4 years
The incidence, character and severity of adverse events as assessed per NCI-CTCAE v5.0 criteria | Through study completion, an average of 4 years
The maximum plasma concentration observed (Cmax) | Through study completion, an average of 4 years
Time of maximum observed plasma concentration (Tmax) | Through study completion, an average of 4 years
Elimination half-life (t1/2) | Through study completion, an average of 4 years
AUC0-∞ | Through study completion, an average of 4 years
AUC0-t | Through study completion, an average of 4 years
Apparent clearance (CL/F) | Through study completion, an average of 4 years
Apparent volume of distribution (Vz/F) | Through study completion, an average of 4 years

OTHER OUTCOMES:
Colony-stimulating factor (CSF) concentrations | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No